CLINICAL TRIAL: NCT01083992
Title: Role of Vitagliptin and Vitamin D in the Treatment of Non Alcoholic Fatty Liver Disease (NAFLD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Liver Clinic, Ziv medical center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAFLD+ Vitamin D
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2010-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: NAFLD; Galvus; vitamin D
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Vildagliptin; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Galvus + vitamin D (Other): Galvus in combination with vitamin D
  Interventions: Drug: Galvus + vitamin D
- Galvus (Other): vitagliptin as monotherapy
  Interventions: Drug: Galvus (vitagliptin)

INTERVENTIONS:
Drug: Galvus (vitagliptin) — Galvus (vitagliptin)
  Arms: Galvus
Drug: Galvus + vitamin D — Galvus + vitamin D
  Arms: Galvus + vitamin D

SUMMARY:
Sedentary lifestyle and poor dietary choices are leading to a weight gain epidemic and increasing the risk for developing nonalcoholic fatty liver disease (NAFLD). The strong relationship between insulin resistance and NAFLD suggests that adding Vitamin D TO insulin sensitizing therapies such as Galvus (vitagliptin) might be beneficial in the prevention or improvement in NAFLD. Considering the close relationship between NAFLD and T2DM and lipid metabolism, we assume that adding vitamin D to Galvus, may be effective for NAFLD by improving lipid metabolism and by improving type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
Sedentary lifestyle and poor dietary choices are leading to a weight gain epidemic and increasing the risk for developing nonalcoholic fatty liver disease (NAFLD). The strong relationship between insulin resistance and NAFLD suggests that adding vitamin D to insulin sensitizing therapies such as Galvus (vitagliptin) might be beneficial in the prevention or improvement in NAFLD. Considering the close relationship between NAFLD and T2DM and lipid metabolism, we assume that adding vitamin D to Galvus may be effective for NAFLD by improving lipid metabolism and by improving T2DM. Methods: 60 patients with NAFLD (Diagnosed by Ultrasound, increase ALT level and hepatomegaly) will be enrolled, and divided into 2 arms Galvus plus Vitamin D vs. Galvus alone. Biochemistry, hepatic triglycerides, histology, m RNA gene expression of collagen, MTP, SREP-1, PPAR-alpha, and LDLR will be measured. 2 separate liver biopsies will be performed at screening and 6 months from baseline. Expected results: Long-term combination therapy with vitagliptin and Vitamin D significantly reduced steatosis, inflammation and fibrosis in the liver compared with long-term monotherapy. We expect also that the combination therapy also significantly increased the expression of microsomal triglyceride transfer protein (MTP) and peroxisome proliferators-activated receptor-α1 (PPAR-α1) in the liver, compared with monotherapy, which may have lead to the improvement in lipid metabolic disorder . Conclusion: Combination therapy of vitagliptin and vitamin D, for 24 weeks improve the histopathology findings in NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Men and women with NAFLD per US
* Increased ALT level
* Hepatomegaly
* Liver biopsy within 2 years

Exclusion Criteria:

* Other liver diseases (HBV, HCV)
* Hepatocellular carcinoma
* Decompensated liver disease
* Use of steroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-01 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
decrease in histological findings | 6 months
  decrease in histological findings: decrease in fat concentration and fibrosis degree

CONTACTS AND LOCATIONS:
Overall Officials: Nimer Assy, MD, Principal Investigator — ZIV MEDICAL CENTER, SAFED ISRAEL; ASSY NIMER, MD, Principal Investigator — Ziv medical center safed, israel
Locations (1):
- Ziv medical center liver unit, Safed, Israel, Israel